CLINICAL TRIAL: NCT04215718
Title: Fistulotomy With Marsupialization Versus Fistulectomy With Wound Sutures in Simple Anal Fistula, a Comparative Clinical Trial
Brief Title: Fistulotomy With Marsupialization Versus Fistulectomy With Wound Sutures in Simple Anal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anal fistula wound
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Fistula in Ano
Keywords: fistula in ano; fistulectomy wound closure; fistulotomy wound marsupialization
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: 2 groups of patients with simple anal fistula each one 46 patients the1st underwent fistulotomy with marsupialization of wound edges the second underwent fistulectomy and wound closure
Who Masked: Participant
Masking Description: the patients don't know which procedure they underwent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fistulotomy group (Active Comparator): 46 patients with simple anal fistula underwent fistulotomy and marsupialization of wound edges
  Interventions: Procedure: fistulotomy and marsupialization
- fistulectomy group (Active Comparator): 46 patients with simple anal fistula underwent fistulectomy and closure of the wound
  Interventions: Procedure: fistulectomy and wound closure

INTERVENTIONS:
Procedure: fistulotomy and marsupialization — the anal fistula was laid open and the the wound edges was marsupialized using vicryle 3\0 sutures
  Arms: fistulotomy group
Procedure: fistulectomy and wound closure — anal fistula was excised with both openings and the wound was closed
  Arms: fistulectomy group

SUMMARY:
comparison between fistulectomy wound closure and fistulotomw wound marsupialization in treatment of simple anal fistula

DETAILED DESCRIPTION:
the investigators conducted this comparative clinical trial in the period between April 2017 and March 2019, on 92 patients with simple anal fistula, patients were randomly allocated into 2 groups, group I the fistulotomy group; 46 patients they underwent fistulotomy and marsupialization of wound edges. Group II, the fistulectomy group they underwent fistulectomy with closure of the wound.

Randomization was done using computer generated cards, the trial was approved by institutional review board (IRB) and the ethical committee of our hospitals, all study participants signed an informed written consent.

The condition of this trial is simple anal fistula defined as non-branched fistula confined to the lower third of the anal sphincter diagnosed by anorectal examination or MRI if needed, the primary outcomes are; the time taken for complete healing, fistula recurrence and anal incontinence diagnosed by Vaizey score patient's questionnaire. The secondary outcomes are local wound complications and postoperative pain calculated by visual analogue score (VAS). Study participants number was calculated through the IRB depending on the incidence of simple anal fistula in our locality.

inclusion criteria

• patients above 18 years diagnosed with simple non recurrent anal fistula.

exclusion criteria:

* Anorectal malignancy.
* Specific disease (Crohn's disease).
* ASA class III, VI and any contraindication for surgery
* Immunocompromised patients and those on steroid therapy or cytotoxic drugs.
* Perianal collection. participants of this study were subjected to proper history taking and full clinical examination for diagnosis of the condition, detection of any associated disease and \ or exclusion factor. MRI was ordered if there is any doubt about diagnosis, preoperative investigations were ordered as per usual.

The procedure in both groups was carried out by the study surgeons, under general anesthesia in lithotomy position, anorectal examination was done to identify the internal and external openings, course of fistulous track and any side tracks if present. When the internal opening couldn't be identified the operator used methylene blue dye injection through the external opening. In fistulotomy group and after probing of the track it was let open by diathermy, its floor was curetted and the wound edges marsupialized by polygalactin (Vicryl) sutures 3\0.

In fistulectomy group and after probing, the fistulous track was excised by diathermy together with its internal and external openings, after hemostasis the wound was closed by polygalactin (Vicryl) sutures 3\0.

In both groups the wound was dressed with non-adhesive dressing, Nonsteroidal analgesics were given as per need and participants were discharged after 24 hours if there is no contraindication to do so.

After discharge study participants were encouraged for self-cleaning by antiseptic baths.

Follow up was carried out in the outpatient clinics by the study surgeons, the clinic visits were planed every week for 12 weeks then monthly for another three months, in each visit the investigator recorded the state of wound healing, anal continence, postoperative pain, any local wound complications, and any recurrence after complete healing in the follow up time.

Preoperative data, demographic data, operative time, intraoperative complications and follow up data were collected and properly analyzed using paired t test and Z tests in SPSS 22 program package.

ELIGIBILITY:
Inclusion Criteria:

• patients above 18 years diagnosed with simple non recurrent anal fistula.

Exclusion Criteria:

* Anorectal malignancy.
* Specific disease (Crohn's disease).
* ASA class III, VI and any contraindication for surgery
* Immunocompromized patients and those on steroid therapy or cytotoxic drugs.
* Perianal collection.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
healing time | 8 weeks
  time taken for complete epithelialization of the wound detected by clinical examination
number of participants with recurrence of anal fistula | 6 months
  presence of anal fistula after complete wound healing detected by clinical examination
number of participants with anal incontinence | i months
  inability to control stool or flatus diagnosed by Vaizey score questionaire

SECONDARY OUTCOMES:
number of participants with postoperative pain and its degree | 1 week
  degree of postoperative pain detected by visual analogue scale calculation
number of participants with post operative complications | 1 week
  post operative complications as bleeding and wound infection detected by clinical examination
operative time | 1 hour
  time of the procedures calculated in minutes starting with the first incision to the start of wound dressing

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, MD, Principal Investigator — zag university
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: No